CLINICAL TRIAL: NCT03616457
Title: Evaluation of Automated Breast Ultrasound as an Adjunct to Screening Digital Breast Tomosynthesis in Women With Dense Breasts (AMELIA)
Brief Title: Automated Breast Ultrasound as an Adjunct to Screening Digital Breast Tomosynthesis
Acronym: AMELIA
Status: Withdrawn | Type: Observational
Why Stopped: Change in business need.
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: 110.01-2018-GES-0001
Record Dates: First submitted 2018-07-26; First posted 2018-08-06 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Breast Cancer
Keywords: Screening Diagnostic
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- All Study Participants: All study participants will undergo the same study procedures, including Automated Breast Ultrasound (ABUS).
  Interventions: Device: Automated Breast Ultrasound (ABUS)

INTERVENTIONS:
Device: Automated Breast Ultrasound (ABUS) — Participants will undergo imaging with ABUS.

SUMMARY:
The purpose of this study is to assess whether the Invenia™ Automated Breast Ultrasound (ABUS) device, as an adjunct to Digital Breast Tomosynthesis (DBT), improves breast cancer detection in women with dense breasts. The study aims to collect information about cancer detection, treatment, and outcomes based on individual and combined technologies in patients who receive ABUS exams in addition to DBT. The results of this study are intended to be used to extend understanding of ABUS as an adjunct in DBT screening in patients with dense breasts.

DETAILED DESCRIPTION:
Following consenting procedures, subjects will undergo standard of care DBT of both breasts or of one breast if they have had prior uni-lateral mastectomy. Subjects will also undergo ABUS of both breasts or of one breast if they have had prior uni-lateral mastectomy. These imaging exams will be done per the sites routine practice, and can be done in any order.

Images will be read and assessed by one (1) Mammography Quality Standards Act (MQSA)-qualified reader. The evaluating radiologist will use the image reconstruction views appropriate for the evaluation, per his or her medical judgment, and handle diagnostic evaluations in accordance with the standard of care at the investigational site. The DBT images will be read and assessed first and independent of ABUS images. DBT plus ABUS will then be read per routine practice and assessed. Images will not be read until both imaging exams have been completed.

If screening shows a suspicious finding, subjects will receive standard of care follow-up and appropriate workup, which may include biopsy (as needed), to determine cancer status. Subjects will be followed at approximately one year (11- to 16-months) unless negative histopathology with image concordance or positive cancer status is histologically determined prior to one-year follow-up. Follow up procedures will be conducted as per the sites standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Are asymptomatic adult women (aged 40 years or older);
2. Are presenting for a DBT breast cancer screening exam;
3. Have heterogeneously dense or extremely dense breasts (BI-RADS C or D)
4. Are able and willing to participate.

Exclusion Criteria:

1. Have been previously included in this study;
2. Have undergone diagnostic or surgical intervention in the last 12 months, including, but not limited to, core or open biopsy, clip placement, fine-needle aspiration, cytopunction, breast reduction or reconstruction, implant removals; OR
3. Have had a breast cancer diagnosis or treatment in the past 12 months and have re-entered the screening population.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: This study will enroll asymptomatic adults who are clinically referred for breast cancer screening. Participants in this study will be representative of the clinical population.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-08 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Cancer Detection Rate | up to 16 months
  Cancer detection rate of DBT plus ABUS and DBT alone

SECONDARY OUTCOMES:
Invasive Cancer Detection | up to 16 months
  To demonstrate DBT plus ABUS has non-inferior invasive cancer detection relative to DBT alone in women with dense breasts
Positive Predictive Value | up to 16 months
  To demonstrate DBT plus ABUS has non-inferior positive predictive value (PPV 1) for breast cancer relative to DBT alone in women with dense breasts.
Recall Rates | up to 16 months
  To summarize recall rate of DBT plus ABUS in relation to the recall rate of DBT alone for breast cancer screening in dense breasts.

CONTACTS AND LOCATIONS:
Overall Officials: Georgia Spear, Principal Investigator — Endeavor Health